CLINICAL TRIAL: NCT01669993
Title: Factors Predictive of Adverse Postoperative Outcomes in Children Undergoing
Brief Title: Factors Predictive of Adverse Postoperative Outcomes in Children Undergoing Tonsillectomy
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0273
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Tonsillectomy Postoperative Adverse Events
Keywords: Outcomes; Quality improvement; Patient Safety; PACU; Complications; Adverse events; Respiratory arrest; Pain; PONV; Age; Neonate; Infant; Child; Ambulatory; Inpatient; General Anesthesia; Otolaryngology; Tonsillectomy; Obstructive sleep apnea
MeSH Terms: conditions — Apnea; Pain; Postoperative Nausea and Vomiting; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of the study are to identify 1) the patient (demographic and clinical) and health care system factors predictive of immediate and late postoperative adverse outcomes in children undergoing tonsillectomy. 2) Evaluate the preoperative use of the sleep questionnaire to identify children at risk for immediate and late postoperative adverse outcomes in children undergoing tonsillectomy.

DETAILED DESCRIPTION:
Currently, children are scheduled to go home or stay in the hospital depending on expert consensus and institutional guidelines. The investigators preliminary experience (Dr. Sadhasivam PI: IRB No. 2008-0848) with the pharmocogenetic study, studying the phenotypic and genotypic influences of pain and use of opioids in patients undergoing tonsillectomy indicates that a significant number of patients scheduled as outpatients experience prolonged recovery phases in the PACU, some of whom are admitted or re-admitted following discharge. The identification of those factors that are, predictive of adverse events in tonsillectomy patients and the development of a prototype prediction model in this single-center study to support clinical decision-making. The rationale of this project is that developing a model to predict postoperative adverse events will not only lead to improved clinical outcomes and enhance patient safety, but also reduce family psychosocial distress associated with unanticipated hospital visits or re-admission, while reducing the burden on the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-17 years of age
* Children scheduled for tonsillectomy or adeno-tonsillectomy
* ASA I, II, or III

Exclusion Criteria:

* ASA IV and V

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing adenotonsillectomy in the United States
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2012-05; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Emergency Room Admissions | Upto 3 weeks after surgery

SECONDARY OUTCOMES:
Postoperative Adverse Event | Assessed in post anesthesia care unit
  This will be measured in post anesthesia care unit (PACU) and will be a composite measure of any one or a combination of these: desaturation, somnolence, laryngospasm /airway obstruction, airway instrumentation, drug administration, PACU discharge criteria not met, unanticipated hospital or ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Subramanyam, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Jaryszak EM, Lander L, Patel AK, Choi SS, Shah RK. Prolonged recovery after out-patient pediatric adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2011 Apr;75(4):585-8. doi: 10.1016/j.ijporl.2011.01.024. Epub 2011 Feb 15. PMID 21324535
- [Background] Bhattacharyya N, Lin HW. Changes and consistencies in the epidemiology of pediatric adenotonsillar surgery, 1996-2006. Otolaryngol Head Neck Surg. 2010 Nov;143(5):680-4. doi: 10.1016/j.otohns.2010.06.918. PMID 20974339
- [Background] Morris LG, Lieberman SM, Reitzen SD, Edelstein DR, Ziff DJ, Katz A, Komisar A. Characteristics and outcomes of malpractice claims after tonsillectomy. Otolaryngol Head Neck Surg. 2008 Mar;138(3):315-20. doi: 10.1016/j.otohns.2007.11.024. PMID 18312878
- [Background] Stevenson AN, Myer CM 3rd, Shuler MD, Singer PS. Complications and legal outcomes of tonsillectomy malpractice claims. Laryngoscope. 2012 Jan;122(1):71-4. doi: 10.1002/lary.22438. Epub 2011 Nov 10. PMID 22076638
- [Background] Richmond KH, Wetmore RF, Baranak CC. Postoperative complications following tonsillectomy and adenoidectomy--who is at risk? Int J Pediatr Otorhinolaryngol. 1987 Aug;13(2):117-24. doi: 10.1016/0165-5876(87)90088-7. PMID 3667091
- [Background] Raghavendran S, Bagry H, Detheux G, Zhang X, Brouillette RT, Brown KA. An anesthetic management protocol to decrease respiratory complications after adenotonsillectomy in children with severe sleep apnea. Anesth Analg. 2010 Apr 1;110(4):1093-101. doi: 10.1213/ANE.0b013e3181cfc435. Epub 2010 Feb 8. PMID 20142343
- [Background] Brown KA. Outcome, risk, and error and the child with obstructive sleep apnea. Paediatr Anaesth. 2011 Jul;21(7):771-80. doi: 10.1111/j.1460-9592.2011.03597.x. Epub 2011 May 3. PMID 21539679
- [Background] Boss EF, Marsteller JA, Simon AE. Outpatient tonsillectomy in children: demographic and geographic variation in the United States, 2006. J Pediatr. 2012 May;160(5):814-9. doi: 10.1016/j.jpeds.2011.11.041. Epub 2011 Dec 17. PMID 22183449
- [Background] Chervin RD, Hedger K, Dillon JE, Pituch KJ. Pediatric sleep questionnaire (PSQ): validity and reliability of scales for sleep-disordered breathing, snoring, sleepiness, and behavioral problems. Sleep Med. 2000 Feb 1;1(1):21-32. doi: 10.1016/s1389-9457(99)00009-x. PMID 10733617
- [Background] Audit NP. Impact of NICE guidance on rates of haemorrhage after tonsillectomy: an evaluation of guidance issued during an ongoing national tonsillectomy audit. Qual Saf Health Care. 2008 Aug;17(4):264-8. doi: 10.1136/qshc.2006.021386. PMID 18678723
- [Background] Zhao YC, Berkowitz RG. Prolonged hospitalization following tonsillectomy in healthy children. Int J Pediatr Otorhinolaryngol. 2006 Nov;70(11):1885-9. doi: 10.1016/j.ijporl.2006.06.015. Epub 2006 Aug 17. PMID 16919338
- [Background] Mitchell RB, Kelly J. Behavior, neurocognition and quality-of-life in children with sleep-disordered breathing. Int J Pediatr Otorhinolaryngol. 2006 Mar;70(3):395-406. doi: 10.1016/j.ijporl.2005.10.020. PMID 16321451
- [Background] Tunkel DE. Polysomnography before tonsillectomy in children: who and when? Otolaryngol Head Neck Surg. 2012 Feb;146(2):191-3; discussion 194-5. doi: 10.1177/0194599811429236. Epub 2011 Nov 16. PMID 22095954
- [Background] Chervin RD, Weatherly RA, Garetz SL, Ruzicka DL, Giordani BJ, Hodges EK, Dillon JE, Guire KE. Pediatric sleep questionnaire: prediction of sleep apnea and outcomes. Arch Otolaryngol Head Neck Surg. 2007 Mar;133(3):216-22. doi: 10.1001/archotol.133.3.216. PMID 17372077
- [Background] Shapiro NL, Seid AB, Pransky SM, Kearns DB, Magit AE, Silva P. Adenotonsillectomy in the very young patient: cost analysis of two methods of postoperative care. Int J Pediatr Otorhinolaryngol. 1999 May 5;48(2):109-15. doi: 10.1016/s0165-5876(99)00011-7. PMID 10375035
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Varughese AM, Morillo-Delerme J, Kurth CD. Quality management in the delivery of pediatric anesthesia care. Int Anesthesiol Clin. 2006 Winter;44(1):119-39. doi: 10.1097/01.aia.0000196253.46033.f9. No abstract available. PMID 16394837
- [Background] Varughese AM, Nick TG, Gunter J, Wang Y, Kurth CD. Factors predictive of poor behavioral compliance during inhaled induction in children. Anesth Analg. 2008 Aug;107(2):413-21. doi: 10.1213/ane.0b013e31817e616b. PMID 18633018
- [Background] Brigger MT, Brietzke SE. Outpatient tonsillectomy in children: a systematic review. Otolaryngol Head Neck Surg. 2006 Jul;135(1):1-7. doi: 10.1016/j.otohns.2006.02.036. PMID 16815173
- [Background] Raeder J. Ambulatory anesthesia aspects for tonsillectomy and abrasion in children. Curr Opin Anaesthesiol. 2011 Dec;24(6):620-6. doi: 10.1097/ACO.0b013e32834b9482. PMID 21897214
- [Background] Sadhasivam S, Chidambaran V, Ngamprasertwong P, Esslinger HR, Prows C, Zhang X, Martin LJ, McAuliffe J. Race and unequal burden of perioperative pain and opioid related adverse effects in children. Pediatrics. 2012 May;129(5):832-8. doi: 10.1542/peds.2011-2607. Epub 2012 Apr 23. PMID 22529273
- [Derived] Subramanyam R, Willging P, Ding L, Yang G, Varughese A. Factors Associated With Postadenotonsillectomy Unexpected Admissions in Children. Anesth Analg. 2021 Jun 1;132(6):1700-1709. doi: 10.1213/ANE.0000000000005123. PMID 32833717